CLINICAL TRIAL: NCT03755362
Title: Treatment of Periodontitis to Prevent Dementia in Older Adults With Asymptomatic Carotid Artery Stenosis and Mild Cognitive Impairment
Brief Title: Dental Carotid Cognitive Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The COVID-19 pandemic has disrupted our ability to continue this study. Follow-up visits were missed to the COVID-19 pandemic restrictions. We have elected to close enrollment and stop follow-up visits.
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: University of Maryland, College Park (Other); Baltimore VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Brajesh Lal, Study Principal Investigator, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HP-00082777
Record Dates: First submitted 2018-11-12; First posted 2018-11-28 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Carotid Stenosis; Mild Cognitive Impairment; Periodontitis
Keywords: carotid stenosis cognitive function periodontitis
MeSH Terms: conditions — Carotid Stenosis; Cognitive Dysfunction; Periodontitis

STUDY DESIGN:
Intervention Model Description: This study will randomize 60 subjects ≥65 years old with asymptomatic carotid artery stenosis (ACAS), mild to moderate cognitive impairment and periodontitis. These 60 patients will be randomized to two groups (intensive vs. standardized periodontal treatment). As randomization will be computer generated, the likelihood of randomization to either group is 50:50.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard treatment (control) (Active Comparator): Dental evaluation and dental prophylaxis at baseline, 3, 6, and 9 months and standard oral hygiene instruction.
  Interventions: Procedure: Standard Treatment
- Intensive Treatment (Experimental): Dental evaluation at baseline, 3, 6, and 9 months. Plus one or more sessions as needed at baseline of full mouth supra- and sub-gingival scaling and root planing, plus oral hygiene instruction. Additional sessions as necessary to remove remaining local factors and treat inflammation and bacteria overgrowth. Additional evaluations and therapy at 2 months or as needed based on therapeutic response. If bleeding on probing levels do not decrease to <20% of sites following initial therapy or at subsequent visits, intermediate treatment visits will be scheduled. Each participant will be instructed to use half of a capful of 0.12% chlorhexidine twice a day during active treatment including two weeks beyond the treatment visit.
  Interventions: Procedure: Intensive Treatment

INTERVENTIONS:
Procedure: Standard Treatment — Dental evaluation at baseline, 3, 6, and 9 months.
  Arms: Standard treatment (control)
Procedure: Intensive Treatment — Dental evaluation at baseline, 3, 6, and 9 months. Plus one or more sessions as needed at baseline of full mouth supra- and sub-gingival scaling and root planing, plus oral hygiene instruction. Additional sessions as necessary to remove remaining local factors and treat inflammation and bacteria overgrowth. Additional evaluations and therapy at 2 months or as needed based on therapeutic response. If bleeding on probing levels do not decrease to <20% of sites following initial therapy or at subsequent visits, intermediate treatment visits will be scheduled. Each participant will be instructed to use half of a capful of 0.12% chlorhexidine twice a day during active treatment including two weeks beyond the treatment visit.
  Arms: Intensive Treatment

SUMMARY:
Periodontal Disease (PD) is present in 60+% of adults >65 years and is associated with tobacco smoking, diabetes, and atherosclerosis that worsen inflammation, comorbidities common in older people with mild to moderate cognitive impairment (MCI). Older MCI patients are prone to poor oral hygiene and dental health, which if untreated worsens inflammation-mediated brain and nervous system function, and accelerates progression to dementia. Asymptomatic carotid artery stenosis (ACAS) is often a silent disease detected in only ~10% of older adults, and may have a strong association with MCI. This study examines the effects of intensive therapy for periodontitis on cognition in high-risk older people with ACAS. Results could highlight PD as a readily modifiable risk factor for dementia.

DETAILED DESCRIPTION:
Periodontal Disease (PD) is present in 60+% of adults >65 years and is associated with tobacco smoking, diabetes, and atherosclerosis that worsen inflammation, comorbidities common in older people with mild to moderate cognitive impairment (MCI). Older MCI patients are prone to poor oral hygiene and dental health, which if untreated worsens inflammation-mediated brain and nervous system function, and accelerates progression to dementia. Asymptomatic carotid artery stenosis (ACAS) is often a silent disease detected in only ~10% of older adults, and may have a strong association with MCI. This study examines the effects of intensive therapy for periodontitis on cognition in high-risk older people with ACAS. Results could highlight PD as a readily modifiable risk factor for dementia.

This pilot study examines the hypothesis that intensive treatment of PD (IPT) in older people with MCI and ACAS will attenuate their cognitive decline by reducing oral microbial-mediated inflammation and improving cerebrovascular endothelial function that contribute to neurodegeneration-associated dementia.

The aims are to determine the effects of intensive compared to control PD treatment (randomized: IPT vs. CPT) in 60 MCI subjects with ACAS and PD on 1) Cognitive function (Primary Outcome) and quality of life (Secondary Outcome), and 2) The potential mechanisms mediating these effects

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or greater than 65 years.
* Body Mass Index 18-35 kg/m2
* Mild to moderate periodontitis
* Mild to moderate cognitive impairment on Montreal Cognitive Assessment (MoCA) -range greater than or equal to 17 and less than or equal to 26 (i.e., range from 17-26).
* Detectable carotid plaque and carotid artery stenosis <70% as diagnosed by doppler ultrasound.
* Able to perform prescribed dental hygiene and travel to medical center as required to participate in the study.

Exclusion Criteria:

* Inability to provide informed consent.
* Subjects with inability to perform cognitive and other research testing
* Prior stroke, depression (CESD >16), neurologic or psychiatric disease that would affect cognitive testing, participation, and compliance to the research study.
* Subjects requiring chronic treatment with systemic corticosteroids or other systemic immunosuppressive drugs or drugs that would affect the dental treatments in the protocol are excluded.
* Subjects requiring essential dental care (e.g., treatment for grossly decayed teeth, broken teeth, dental abscesses, peri-apical infections, other dental infections).
* Inability to perform FDG-PET due to renal disease (eGFR <30 mL/min/1.75m2).
* Receiving anticoagulant therapy (Warfarin) with an INR greater than 3.3 at time of dental treatment or with a bleeding disorder, or other diseases that may interfere with dental therapy.
* Subjects with medical conditions that the clinicians feel would limit their ability to participate.

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2021-02-21 (Actual); Study Completion 2021-02-25 (Actual)

PRIMARY OUTCOMES:
Changes in performance on Montreal Cognitive Assessment (MoCA) | 1 year
  The Montreal Cognitive Assessment (MoCA) is 30 item screening tool used to detect cognitive impairment. Score: 30 points (maximum), 0 points (minimum). Higher scores indicate better cognitive function. Differences in rate of change of MoCA score in those on intensive treatment for periodontitis and those receiving standard care.

SECONDARY OUTCOMES:
Presence of oral bacteria in saliva and dental plaque samples | 1 year
  Dental plaque and saliva samples will be analyzed for differences in species of oral microbial biology between those on standard care compared to those on intensive treatment for periodontitis. Oral microbiome will be characterized using molecular genetic methods.
Presence of bacteria in stool samples | 1 year
  Stool samples will be analyzed for differences in species of oral microbial biology between those on standard care compared to those on intensive treatment for periodontitis. Stool microbiome will be characterized using molecular genetic methods.
Systemic inflammation | 1 year
  Differences in inflammatory markers such as Interleukin 6 (IL-6) and tumor necrosis factor (TNF) alpha found in blood samples in those on standard care compared to those on intensive treatment for periodontitis.
Change from baseline in Fluorodeoxyglucose Positron Emission Tomography (FDG-PET) Metabolic Measure of Standard Uptake Value Ratio (SUVR) | 1 year
  Brain metabolic activity or glucose metabolism will be determined using the FDG-PET scan by reporting results as SUVR and compared in those on intensive treatment for periodontitis and those receiving standard treatment for periodontitis.
Changes in performance on Wechsler Adult Intelligence Scale (WAIS)-III Digit Span subtest | 1 year
  Change in Digit Span score as a measure of working memory in those on standard care compared to those on intensive treatment for periodontitis. Raw score: 0-30, t score 19-77
Changes in performance on Hopkins Verbal Learning Test | 1 year
  Change in Hopkins Verbal Learning test score in those on standard care compared to those on intensive treatment for periodontitis. Total raw score: 0 (minimum)-36 (maximum), t score 19-77. Higher scores indicate higher functioning.
Changes in performance on Brief Visuospatial Memory test | 1 year
  Change in Brief Visuospatial Memory test score in those on standard care compared to those on intensive treatment for periodontitis. Total raw score : 0 (minimum)-36 (maximum), t score 19-77. Higher scores indicate higher functioning.
Changes in performance on Trail Making Test (A+B) | 1 year
  Change in Trail Making Test (A+B) score as a measure of visual attention and task switching in those on standard care compared to those on intensive treatment for periodontitis. Range: 10-400 seconds; t score 19-77. Lower times indicate higher functioning.
Changes in performance on Controlled Oral Word Association Test | 1 year
  Change in Controlled Oral Word Association Test as a measure of verbal fluency score in those on standard care compared to those on intensive treatment for periodontitis. Total raw score : 0 (minimum)-90 (maximum); t score 19-77. Higher scores indicate higher functioning.
Changes in performance on Boston Naming Test | 1 year
  Change in Boston Naming Test score as a measure of confrontational word retrieval in those on standard care compared to those on intensive treatment for periodontitis. Total raw score : 0 (minimum)-60 (maximum); t score 19-77. Higher scores indicate higher functioning.
Changes in performance on Modified Wisconsin Card Sorting Test | 1 year
  Change in Modified Wisconsin Card Sorting Test score as a measure of abstract reasoning ability in those on standard care compared to those on intensive treatment for periodontitis. Number of categories score : 0 (minimum)-6(maximum); t score 19-77. Higher scores indicate higher functioning.
Changes in performance on Grooved Pegboard Test | 1 year
  Change in Grooved Pegboard Test score as a measure of visual-motor coordination in those on standard care compared to those on intensive treatment for periodontitis. Range: 10-500 seconds; t score 19-77. Lower times indicate higher functioning.
Changes in Composite Cognitive Function Score | 1 year
  Change in composite cognitive function in those on standard care compared to those on intensive treatment for periodontitis. T scores (19-77) of individual neuropsychological tests will be averaged to compute composite scores. Neuropsychological tests include: Digit span, Hopkins Verbal Learning Test, Brief Visuospatial Memory test, Trail Making Test (A+B), Controlled Oral Word Association Test, Grooved Pegboard Test, Boston Naming Test, Modified Wisconsin Card Sorting Test.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberlly Nordstrom, CCRC, Study Director — University of Maryland, College Park
Locations (1):
- University of Maryland - Administrative Center, Baltimore, Maryland, United States

REFERENCES:
- [Background] Gorelick PB, Scuteri A, Black SE, Decarli C, Greenberg SM, Iadecola C, Launer LJ, Laurent S, Lopez OL, Nyenhuis D, Petersen RC, Schneider JA, Tzourio C, Arnett DK, Bennett DA, Chui HC, Higashida RT, Lindquist R, Nilsson PM, Roman GC, Sellke FW, Seshadri S; American Heart Association Stroke Council, Council on Epidemiology and Prevention, Council on Cardiovascular Nursing, Council on Cardiovascular Radiology and Intervention, and Council on Cardiovascular Surgery and Anesthesia. Vascular contributions to cognitive impairment and dementia: a statement for healthcare professionals from the american heart association/american stroke association. Stroke. 2011 Sep;42(9):2672-713. doi: 10.1161/STR.0b013e3182299496. Epub 2011 Jul 21. PMID 21778438
- [Background] Smith JA, Das A, Ray SK, Banik NL. Role of pro-inflammatory cytokines released from microglia in neurodegenerative diseases. Brain Res Bull. 2012 Jan 4;87(1):10-20. doi: 10.1016/j.brainresbull.2011.10.004. Epub 2011 Oct 18. PMID 22024597
- [Background] Leszek J, Barreto GE, Gasiorowski K, Koutsouraki E, Avila-Rodrigues M, Aliev G. Inflammatory Mechanisms and Oxidative Stress as Key Factors Responsible for Progression of Neurodegeneration: Role of Brain Innate Immune System. CNS Neurol Disord Drug Targets. 2016;15(3):329-36. doi: 10.2174/1871527315666160202125914. PMID 26831258
- [Background] Miklossy J, McGeer PL. Common mechanisms involved in Alzheimer's disease and type 2 diabetes: a key role of chronic bacterial infection and inflammation. Aging (Albany NY). 2016 Apr;8(4):575-88. doi: 10.18632/aging.100921. PMID 26961231
- [Background] Otomo-Corgel J, Pucher JJ, Rethman MP, Reynolds MA. State of the science: chronic periodontitis and systemic health. J Evid Based Dent Pract. 2012 Sep;12(3 Suppl):20-8. doi: 10.1016/S1532-3382(12)70006-4. PMID 23040337
- [Background] Daulatzai MA. Cerebral hypoperfusion and glucose hypometabolism: Key pathophysiological modulators promote neurodegeneration, cognitive impairment, and Alzheimer's disease. J Neurosci Res. 2017 Apr;95(4):943-972. doi: 10.1002/jnr.23777. Epub 2016 Jun 27. PMID 27350397
- [Background] Teixeira FB, Saito MT, Matheus FC, Prediger RD, Yamada ES, Maia CSF, Lima RR. Periodontitis and Alzheimer's Disease: A Possible Comorbidity between Oral Chronic Inflammatory Condition and Neuroinflammation. Front Aging Neurosci. 2017 Oct 10;9:327. doi: 10.3389/fnagi.2017.00327. eCollection 2017. PMID 29085294
- [Background] Fouad A, Mongodin E, Hittle L, et al. Microbiome analysis of oral and atheromatous plaques in atherosclerotic patients. In: IADR General Session and Exhibition. 2014
- [Background] Emery DC, Shoemark DK, Batstone TE, Waterfall CM, Coghill JA, Cerajewska TL, Davies M, West NX, Allen SJ. 16S rRNA Next Generation Sequencing Analysis Shows Bacteria in Alzheimer's Post-Mortem Brain. Front Aging Neurosci. 2017 Jun 20;9:195. doi: 10.3389/fnagi.2017.00195. eCollection 2017. PMID 28676754
- [Background] Caminiti SP, Ballarini T, Sala A, Cerami C, Presotto L, Santangelo R, Fallanca F, Vanoli EG, Gianolli L, Iannaccone S, Magnani G, Perani D; BIOMARKAPD Project. FDG-PET and CSF biomarker accuracy in prediction of conversion to different dementias in a large multicentre MCI cohort. Neuroimage Clin. 2018 Jan 28;18:167-177. doi: 10.1016/j.nicl.2018.01.019. eCollection 2018. PMID 29387532
- [Background] Ide M, Harris M, Stevens A, Sussams R, Hopkins V, Culliford D, Fuller J, Ibbett P, Raybould R, Thomas R, Puenter U, Teeling J, Perry VH, Holmes C. Periodontitis and Cognitive Decline in Alzheimer's Disease. PLoS One. 2016 Mar 10;11(3):e0151081. doi: 10.1371/journal.pone.0151081. eCollection 2016. PMID 26963387